CLINICAL TRIAL: NCT07203495
Title: An Observational Clinical Study on the Spatiotemporal Changes and Prognostic Value of the 18F-FDG PET Neuro-Metabolic Network
Brief Title: Spatiotemporal Dynamics and Prognostic Value of the 18F-FDG PET Neuro-Metabolic Network
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, yujie bai, Attending Physician, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2025-KY-1046
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Lung Diseases; Endocrine Diseases; Gastrointestinal Diseases
Keywords: 18F-FDG PET; Brain-organ axis; Neuro-metabolic network
MeSH Terms: conditions — Lung Diseases; Endocrine System Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Individuals aged 18-75 years who, based on medical history, physical examination, laboratory testing, and imaging assessments, are confirmed to be free of target diseases and related complications. This group may include healthy volunteers or individuals recruited from health check-up populations.
- Disease Group: Patients aged 18-75 years with a confirmed diagnosis of lung, gastrointestinal, or endocrine diseases. Participants with organic brain lesions (e.g., stroke, Alzheimer's disease, Parkinson's disease) or psychiatric disorders (e.g., depression, anxiety, schizophrenia), or other conditions that may affect cerebral metabolism or prognosis, will be excluded.

SUMMARY:
This observational clinical study aims to investigate the spatiotemporal changes of the 18F-FDG PET neuro-metabolic network in patients with lung, gastrointestinal, or endocrine diseases. The study seeks to clarify :

1. the dynamic metabolic alterations of specific brain regions,
2. the spatiotemporal associations between cerebral metabolism and systemic disease progression,
3. the prognostic value of neuro-metabolic parameters. Participants will undergo 18F-FDG PET/CT imaging, clinical assessments, and longitudinal follow-up to evaluate outcomes such as tumor recurrence, metastasis, and survival.

DETAILED DESCRIPTION:
The brain-organ axis, including the brain-lung, brain-heart, brain-gut, and brain-endocrine pathways, has emerged as a critical research field for systemic disease pathophysiology. 18F-FDG PET/CT provides a unique noninvasive tool to quantify neural metabolic activity and to reveal central-peripheral interactions in cross-axis disorders. Previous studies have demonstrated that chronic hypoxia in lung diseases can lead to global cerebral metabolic suppression, with prominent hypometabolism in the frontal cortex and hippocampus, directly correlating with cognitive decline. Similarly, brain-heart axis dysfunction in heart failure is characterized by hypothalamic-amygdala hypermetabolism and hippocampal hypometabolism, linked to higher rehospitalization risk. Inflammatory bowel disease demonstrates abnormal hypermetabolism in the insula and anterior cingulate cortex, correlated with intestinal mucosal damage. Moreover, 18F-FDG PET can sensitively detect pituitary microadenomas and predict postoperative recurrence in Cushing's disease.

Despite these advances, three major limitations remain:

1. most studies focus on single organ axes, lacking integrative dynamic network analyses across multiple axes;
2. conventional static SUV metrics cannot capture the spatiotemporal evolution of metabolic pathways, while advanced dynamic PET approaches remain underutilized in clinical practice;
3. prognostic models often rely on single-modality parameters, ignoring the added value of multimodal integration, as shown by recent evidence combining DWI-derived ADC values with PET metabolic parameters to enhance prognostic accuracy in NSCLC.

Therefore, this prospective cohort study will systematically map neuro-metabolic remodeling patterns of brain-organ axis diseases using 18F-FDG PET imaging, and establish metabolism-based prognostic stratification models.

Objectives:

To characterize the dynamic cerebral metabolic alterations in patients with lung, gastrointestinal, or endocrine diseases.

To explore the spatiotemporal associations between specific brain region metabolism and disease progression.

To assess the prognostic value of cerebral metabolic parameters for clinical outcomes.

Primary Outcomes:

The primary outcomes include tumor recurrence, metastasis, and death. All events will be adjudicated by at least two independent clinicians based on comprehensive clinical information and professional expertise. The number and timing of outcome events will be recorded at the end of follow-up for each participant.

ELIGIBILITY:
Inclusion Criteria:

Healthy Control Group: Healthy volunteers or individuals from health check-up populations who, based on medical history, physical examination, laboratory testing, and imaging assessments, are confirmed to be free of target diseases and related complications.

Disease Group: Patients aged 18-75 years with a confirmed diagnosis of lung, gastrointestinal, or endocrine diseases.

Exclusion Criteria:

Presence of organic brain lesions identified on imaging, including but not limited to stroke, Alzheimer's disease (AD), or Parkinson's disease (PD).

History of psychiatric disorders such as depression, anxiety, or schizophrenia, or other conditions that may affect cerebral metabolic imaging or prognosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of two groups: a healthy control group and a disease group.
  Healthy Control Group: Healthy volunteers or individuals recruited from health check-up populations, aged 18-75 years, who are confirmed through medical history, physical examination, laboratory tests, and imaging evaluations to be free of the target diseases and related complications.
  Disease Group: Patients aged 18-75 years with a confirmed diagnosis of lung, gastrointestinal, or endocrine diseases.
  Participants will be excluded if they present with organic brain lesions detected on imaging (including but not limited to stroke, Alzheimer's disease, or Parkinson's disease), have a history of psychiatric disorders such as depression, anxiety, or schizophrenia, or have other conditions that may interfere with cerebral metabolic imaging or influence prognosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
tumor recurrence, metastasis, and death | June 1, 2025 to September 1, 2028
  The primary outcomes include tumor recurrence, metastasis, and death. All events will be adjudicated by at least two independent clinicians based on comprehensive clinical information and professional expertise. The number and timing of outcome events will be recorded at the end of follow-up for each participant.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data (IPD) will be shared:
  Clinical data: demographics, diagnosis, medical history, laboratory results, follow-up information, and outcome events (tumor recurrence, metastasis, death).
  Imaging-derived data: quantitative 18F-FDG PET parameters (e.g., SUV values, metabolic tumor volume [MTV], kinetic parameters, connectivity measures).
  Processed imaging files: de-identified parametric maps and derived neuro-metabolic connectivity matrices.
  Supporting documents: study protocol, data dictionary, and analysis code used for image preprocessing and statistical modeling.

REFERENCES:
- [Background] Valenza G, Matic Z, Catrambone V. The brain-heart axis: integrative cooperation of neural, mechanical and biochemical pathways. Nat Rev Cardiol. 2025 Aug;22(8):537-550. doi: 10.1038/s41569-025-01140-3. Epub 2025 Mar 3. PMID 40033035
- [Background] Zhong T, Duan Y, Li K, Qiu J, Cheng Z, Lu W. Directional interactions from non-small cell lung cancer to brain glucose metabolism revealed by total-body PET imaging. Eur J Nucl Med Mol Imaging. 2025 Oct;52(12):4467-4476. doi: 10.1007/s00259-025-07324-w. Epub 2025 May 9. PMID 40342105
- [Background] Tricarico P, Chardin D, Martin N, Contu S, Hugonnet F, Otto J, Humbert O. Total metabolic tumor volume on 18F-FDG PET/CT is a game-changer for patients with metastatic lung cancer treated with immunotherapy. J Immunother Cancer. 2024 Apr 22;12(4):e007628. doi: 10.1136/jitc-2023-007628. PMID 38649279
- [Background] Eze C, Schmidt-Hegemann NS, Sawicki LM, Kirchner J, Roengvoraphoj O, Kasmann L, Mittlmeier LM, Kunz WG, Tufman A, Dinkel J, Ricke J, Belka C, Manapov F, Unterrainer M. PET/CT imaging for evaluation of multimodal treatment efficacy and toxicity in advanced NSCLC-current state and future directions. Eur J Nucl Med Mol Imaging. 2021 Nov;48(12):3975-3989. doi: 10.1007/s00259-021-05211-8. Epub 2021 Mar 24. PMID 33760957